CLINICAL TRIAL: NCT02817009
Title: Healthy Families: Transforming Care for Obese Children at NYU Lutheran Family Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-00319
Record Dates: First submitted 2016-03-07; First posted 2016-06-29 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Childhood Obesity
Keywords: Behavioral Health Intervention; Randomized Control Trial; Family Intervention; Nutrition; Weight Management; Multidisciplinary Program
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition Group (No Intervention): This group will go through standard of care and visit the nutritionist on a monthly basis for the three months that they are a part of the study.
- Healthy Families Group (Experimental): Participants and their families will attend a weekly nutrition session, social support session and physical activity session for 12 weeks.
  Interventions: Behavioral: Social Support; Behavioral: Nutrition Session; Behavioral: Physical Activity Session

INTERVENTIONS:
Behavioral: Social Support — The social worker for the parent support group addresses culturally specific questions and adopts culturally acceptable strategies for setting limits and promoting healthy behaviors, engaging the group as a whole and building peer support.
  Arms: Healthy Families Group
Behavioral: Nutrition Session — Nutrition sessions will focus on how to make traditional Latin American foods healthier, including the sharing of recipes and learning what foods to buy in local supermarkets. Home visits by the nutritionist assists with family-centric strategies for healthier eating in their urban Latino households, including those with large extended families.
  Arms: Healthy Families Group
Behavioral: Physical Activity Session — 45 minutes physical activity session to promote healthy behaviors
  Arms: Healthy Families Group

SUMMARY:
Childhood obesity is a contributing factor to health complications such as diabetes, heart disease, high blood pressure, cancer and asthma. It is of particular concern among Hispanic populations in the United States as that group has the fastest growing childhood obesity rate. Nearly two in five Hispanic children ages 2 to 19 are overweight or obese. This program aims to test whether it is beneficial to routinize a multi-disciplinary pediatric weight management program within the highest volume clinic (NYU-LFHC Women, Adolescents and Children), and to add a home-visit component to reinforce teaching on food selection and preparation. The intervention will include 27-hour intervention session which will be distributed into 12-session series over a 3 month period. The program will target Hispanic children between the ages of 9 and 11 with a Body Mass Index (BMI) between the 95th and 99th percentiles. To assess the effectiveness of this program, the investigators propose to conduct a general prospective study using randomized pre-test and post-test control group design with minimal risk for participants.

DETAILED DESCRIPTION:
The proposed intervention will engage pediatricians at NYU Lutheran Family Health Centers (NYU LFHC) and providers at the school-based clinics in referring Hispanic children ages 9-11 years with a BMI between the 95th and 99th percentile to the study. In addition, a list will be generated from NYU Lutheran's Quality Improvement department if recruitment through providers is low. Providers will refer patients who meet the above criteria through eClincialWorks (ECW). A research assistant will then randomize the referrals after acquiring informed consent forms to either the control group or the intervention group. The control group will receive standard of care by nutritionists at NYU LFHC. The intervention group will receive a 27-hour intervention session which will be split into a 12-session series. The sessions will be conducted weekly over a 3 month period. This study will include three cycles with three separate cohorts.

The Healthy Families Intervention Group will include:

1. Bilingual English and Spanish group nutrition education, behavioral social support, and physical activity (e.g. kickboxing, Zumba, yoga, aerobics).
2. Monthly home visits by a nutritionist for family including specific recommendations on food purchasing and preparation.

Children randomized to standard of care will attend monthly sessions with a nutritionist.

ELIGIBILITY:
Inclusion Criteria:

* Patient of NYU-LFHC Women's, Pediatric, and Adolescent Medicine (5610)
* Hispanic ethnicity
* BMI percentile between the 95th and 99th
* Ages between 9 and 11 years old at the time the program begins

Exclusion Criteria:

* Autism Spectrum Disorder (299.0)
* Pervasive Developmental Disorder-Not Otherwise Specified (PDD NOS 299.9) and
* Other PDD (299.8)

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Stabilize Body Mass Index (BMI) | 3 months
  The goal is to stabilize or reduce the participant's BMI at the end of the study. The height and weight of the control group will be measured at baseline and at the end of 3 months. The height and weight of the intervention group will be measured at over 12 sessions within the 3 month time frame. The intervention will be 27 hours in total.

SECONDARY OUTCOMES:
Differences in 5-2-1-0 measures between baseline and post-intervention session | 3 months
  Compare pre-intervention and post-intervention data within the control and intervention group for cases for the following behaviors: physical activity, consumption of fruit and vegetables, sugar-sweetened beverages, and daily screen time (watching TV/YouTube, playing video games, using tablet/phone/mobile device), which will be collected through the 5-2-1-0 validated survey.
Stabilize BMI z-score | 3 months
  The goal is to stabilize BMI z-score by the end of 3 months. The BMI z-score will be calculated using the BMI collected in the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Marisol Gonzalez, MD, Principal Investigator — NYU Lutheran
Locations (1):
- NYU Lutheran Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No